CLINICAL TRIAL: NCT05977387
Title: Pediatric Kidney Transplant
Acronym: PeKiT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-21-PeKiT
Record Dates: First submitted 2022-02-08; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: End Stage Renal Disease; Pediatric ALL; Kidney Transplant; Complications
MeSH Terms: conditions — Kidney Failure, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
End-stage renal disease (ESRD) is a rare disease in children. Renal transplantation (RT) is the treatment of choice for ESRD in the pediatric population. In France, around 100 pediatric kidney transplants are performed each year. The aim was to evaluate the surgical management of TR and the long-term results.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a rare pathology in children, whose gold standard treatment is a kidney transplant. In France, around 100 pediatric kidney transplants are performed every year.

Although the first adult kidney transplants were performed in 1954, pediatric renal transplantation was considered unsafe compared with dialysis, which was preferred. In the 1980s, improved graft selection, optimized pre-transplant management and a better understanding of the immune system led to the development of pediatric kidney transplantation.

Despite considerable progress, graft survival in these long-lived patients remains a major challenge.

The aim of this study is to evaluate surgical practices in the four French pediatric transplant centers, and to define risk factors for surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients who underwent renal transplantation in one of the 4 centers

Exclusion Criteria:

* Multi organ transplant

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients from 0 to 18 years who underwent renal transplant for ESRD
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Surgical outcomes | 10 years
  To assess surgical outcome in pediatric renal transplantation in terms of
  * per operative complications (ClassIntra classification)
  * post operative complications (Clavien Dindo) early < 30 days and late > 30 days

SECONDARY OUTCOMES:
Surgical complications | 10 years
  Evaluate the surgical morbidity of renal transplantation
Graft Survival | 10 years
  Evaluate graft survival at 1, 5 and 10 years post transplantation
Return to dialysis | 10 years
  Evaluation of the need to return to dialysis after transplantation : causes and reasons
Retransplantation | 10 years
  Evaluation the number of patient undegoing another transplantation
Death | 10 years
  Evaluation of the morbidity of this population

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - l'hôpital mère-enfant de Lyon, Bron
  - l'hôpital mère enfant de Nantes, Nantes
  - l'hôpital Robert Debré, Paris
  - l'hôpital Necker Enfants malades., Paris